CLINICAL TRIAL: NCT06811233
Title: Monitoring, Detoxifying, and Rebalancing Metals During Acute Myeloid Leukemia (AML) Therapy, a Phase 2 Randomized Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-1369; NCI-2025-00860 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Succimer; Magnesium Sulfate; Geritol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Metal Detoxification with DMSA + Ca-EDTA with Standard AML Therapy (Experimental): Participants treatment will be administered on either an inpatient or outpatient basis
  Interventions: Drug: DMSA; Drug: Ca-EDTA; Drug: Magnesium Sulfate; Drug: Multivitamin

INTERVENTIONS:
Drug: DMSA — Given PO
Drug: Ca-EDTA — Given by IV
Drug: Magnesium Sulfate — Given by infusion
Drug: Multivitamin — Given PO

SUMMARY:
The goal of this clinical research study is to learn if metal detoxification (with calcium disodium edetate [Ca-EDTA] and dimercaptosuccinic acid [DMSA]) during standard therapy can help improve outcomes in patients with intermediate-risk, high-risk, or secondary AML compared to standard therapy alone. Researchers think lowering the level of metals found in the blood/bone marrow may help to control the disease and/or improve the response to chemotherapy.

DETAILED DESCRIPTION:
Primary Objective:

To compare event free survival of patients with newly diagnosed (or untreated) secondary, intermediate, and high-risk AML or newly diagnosed MPN-BP (including CML-BP) receiving metal detoxification during standard therapy to patients with newly diagnosed (or untreated) secondary, intermediate, and high-risk AML or newly diagnosed MPN-BP (including CML-BP) receiving standard therapy alone.

Secondary Objectives:

Compare the remission rates and overall survival rates of patients with newly diagnosed (or untreated) secondary, intermediate, and high-risk AML and newly diagnosed MPN-BP (including CML-BP) receiving metal detoxification during standard therapy to those receiving standard therapy alone.

* To assess the efficacy information regarding the combined therapy in terms of the overall response rate (ORR) including CR, CRh, CRi, MLFS, and PR in patients with newly diagnosed (or untreated) secondary, intermediate, and high-risk AML and newly diagnosed MPN-BP (including CML-BP) receiving metal detoxification during standard therapy and in patients with secondary, intermediate and high-risk AML and newly diagnosed MPN-BP (including CML-BP) receiving standard therapy alone.
* To compare adverse events of patients with newly diagnosed (or untreated) secondary, intermediate, and high-risk AML and newly diagnosed MPN-BP (including CML-BP) receiving metal detoxification during standard therapy to patients with newly diagnosed (or untreated), secondary, intermediate, and high-risk AML and newly diagnosed MPN-BP (including CML-BP) receiving standard therapy alone.
* To assess the complete remission (CR), complete remission with incomplete hematologic recovery (CRi), Complete Remission with Partial hematological recovery (CRh), partial remission (PR), hematologic improvement (HI), morphologic leukemia free state (MLFS) rates, and the overall survival (OS) in AML and MPN-BP patients undergoing cancer therapy combined with DMSA and Ca-EDTA and in patients receiving cancer therapy alone.
* To assess overall survival and event free survival in AML and MPN-BP patients undergoing cancer therapy combined with DMSA and Ca-EDTA and in patients receiving AML therapy alone To assess remission duration in AML and MPN-BP patients undergoing cancer therapy combined with DMSA and Ca-EDTA and in patients receiving AML therapy alone.
* To monitor toxic and essential metal levels during AML therapy combined with DMSA and Ca-EDTA and to evaluate the reduction in metals in the bone marrow and blood of newly diagnosed AML patients undergoing metal detoxification combined with standard AML therapy.
* Correlate metal and copper isotopic abundance ratios of AML patients with clinical data, conventional cytogenetics, extensive Next Generation Sequencing (NGS) (300-gene panel), exposure survey data, and clinical outcome data, and to perform a larger analysis by pooling this data with metal/genomic/survey/outcome data obtained on 2017-0752, 2017-0937 and PA15-0302.
* To assess other responses of interest in Measurement of Effect Section

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent form for participants 18 years or older, unless LAR signs where applicable along with any required verbal assents if patients can provide assent.
2. Age 18 years or older at the time of signing the informed consent form.
3. Diagnosis of Any of the Following:

   * Newly diagnosed (or untreated) AML or Newly diagnosed Myeloproliferative Neoplasm in Myeloid Blast Phase (MPN-BP) [including Chronic Myeloid Leukemia in Blast Phase (CML-BP)], Ph+AML with intermediate-risk or high-risk (by ELN), or any other intermediate or high-risk AML by ELN
   * Secondary AML regardless of ELN risk status, however, may not have CBF [t(8;21) or inv(16)]

   Secondary AML types include:
   * Secondary AML evolved from prior untreated MDS, myeloproliferative neoplasm (MPN), or Aplastic Anemia
   * Therapy-related AML (t-AML)
   * AML evolved after prior MDS, MPN, or Aplastic Anemia after prior therapy for those myeloid bone marrow disorders
   * Secondary AML, including blast phase of MPN (MPN-BP) [also, including CML in blast phase (BP of CML) after prior hematologic myeloid bone marrow disease (MDS, MPN, Aplastic Anemia, CML) (patients may have received treatment for their prior hematologic disorder for their previous bone marrow disorder) . Newly diagnosed (or untreated) myeloid blast phase of MPN (including myeloid blast phase of CML)/Ph+AML.150
4. Patients can enroll on this study after start of non-investigational induction therapy but must be within first 2 cycles of front-line therapy, as long as not in a complete remission.
5. Transformed and untreated AML transformed from previously treated MDS, myeloproliferative neoplasm (MPN) or other types of secondary AML are allowed. Myeloid-Blast Phase of MPN and Myeloid Blast Phase of Chronic Myeloid Leukemia (CML) are allowed/Ph+ AML are allowed.
6. Eastern Cooperative Oncology Group (ECOG) performance status of . 2
7. Laboratory test results within these ranges (unless due to leukemia or other hematologic malignancy):

   * Serum creatinine.2.0 mg/dL
   * Total Bilirubin . 2.0 x Upper limit of normal (ULN) unless the patient has Gilbert fs.
   * AST (SGOT) and/or ALT (SGPT) . 2.0 x ULN
8. Women of childbearing potential (WCBP) must have a negative urine or serum pregnancy test within 14 days and must either commit to continued abstinence from heterosexual intercourse or adopting at least one highly effective method of contraception. These methods include intra-uterine device, tubal ligation, partners vasectomy, and hormonal birth control pills. Men must agree not to father a child and agree to use a condom if his partner is of childbearing potential.
9. Extramedullary disease is allowed if it can be measured and followed for response.

Exclusion Criteria:

1. Nursing and pregnant individuals. Should a study participant become pregnant or suspect pregnancy while participating in this study, the study participant should inform their treating physician immediately.
2. Uncontrolled inter-current illness including, but not limited to, uncontrolled active infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements or which judged by the investigator, places the patient at unacceptable risk.
3. Acute Promyelocytic leukemia (APL)
4. Prior venetoclax failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2031-08-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Maro Ohanian, DO, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org